CLINICAL TRIAL: NCT01672723
Title: Neuropharmacological Basis of Social Connection: The Role of Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Naomi Eisenberger, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Opioids and Social Cognition
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Psychology, Social
Keywords: opioids; social connection
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Experimental): Participants will take 4 doses of naltrexone over 4 days (25mg/day for days 1 and 2, 50mg/day for days 3 and 4) as well as 4 matched placebo pills for a total of 8 days. Capsules will be packaged into blister packs.
  Participants will be asked to take the first drug, either naltrexone or placebo, once a day for three days prior to the first experimental session and when they arrive at the lab for the experimental procedure . After the first session, participants will take the second study drug for three days prior to the second experimental session and when they arrive for the second experimental procedure.
  Interventions: Drug: Naltrexone
- Placebi (Placebo Comparator): Participants will take 4 doses of naltrexone over 4 days (25mg/day for days 1 and 2, 50mg/day for days 3 and 4) as well as 4 matched placebo pills for a total of 8 days. Capsules will be packaged into blister packs.
  Participants will be asked to take the first drug, either naltrexone or placebo, once a day for three days prior to the first experimental session and when they arrive at the lab for the experimental procedure . After the first session, participants will take the second study drug for three days prior to the second experimental session and when they arrive for the second experimental procedure.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone
  Other Names: Depade; ReVia

SUMMARY:
From birth we rely on others for comfort and care and derive pleasure from being together. Research from the fields of health psychology, social psychology, and public health converge to highlight the importance of having and maintaining good relationships for overall health. Indeed, having close friends and family and feeling connected to them has been called a basic need, similar to our need for food and water. It may not be a coincidence then that feelings of connection rely on similar systems in the body as other needs that are both basic and highly pleasing and rewarding. For instance, its possible that opioids, a substance in the body associated with pleasant, euphoric feelings, may also be important for connecting with others. This study will examine the role of opioids in feeling connected to others by administering a drug called naltrexone, that effects opioid processing in the body, on perceptions and feelings toward a number of tasks in the lab. Additionally, to assess the effects of naltrexone outside of the lab, participants will complete daily diary responses via text and online surveys.

40 participants will take both placebo and naltrexone. Participants will complete two sessions, one in each drug condition, in which they complete a number of tasks including reading messages on a computer screen, holding a number of objects, and viewing images while undergoing electric shocks. Participants will also complete a daily diary for 14 days while on naltrexone and placebo. Prior to these lab sessions participants will be screened at UCLA's Clinical & Translational Research Center (CTRC) to ensure that they are healthy and that it is safe for them to take the study drug.

We hypothesize that people will report feeling less socially connected when on naltrexone compared to placebo and will show subsequent changes in social behavior outside of the lab.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the study require that participants be in good health, between the ages of 18 and 35, fluent in English, have access to text messaging technology, and have at least 8 close friends and family members who would be willing to be contacted in regards to the study (for the social connection lab task) and be willing to provide 2 pictures of a close other (for the threat of shock task).

Exclusion Criteria:

Following an email screening and structured telephone interview, prospective participants with the following conditions will not advance to the in- person screening session: pregnant or planning to become pregnant in the next 6 months, presence of chronic mental or physical illness, history of allergies, liver, or other severe chronic diseases, current and regular use of prescription medications, or previous history of fainting during blood draws.

Furthermore, the absence of significant health problems or medication use history will be confirmed by an in-person screening session. Any participant who has any of the following conditions will be ineligible for the study: (1) Any and all medical conditions, especially hepatitis or liver failure.

Psychiatric Disorders. (2) current and/or lifetime history of a major Depressive Disorder or other Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-IV) psychiatric disorder (e.g. substance dependence) (3) current and/or past regular use of analgesics such as opioids; (4) current and/or past regular use of psychotropic medications, including selective serotonergic reuptake inhibitors, antidepressants, anxiolytics, hypnotics, sedatives and barbiturates. Health factors. (5) current smokers (13) body mass index (BMI) greater than 35, (14) shows evidence of drug use from a urine test, (15) has a positive pregnancy test, if female, or (16) shows any abnormalities on screening laboratory tests.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I Eisenberger, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles Department of Psychology, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the UCLA community and surrounding areas and were run between December 2012 and February 2014.
Pre-assignment Details: 50 screened, 19 excluded (1 asked to be removed, 15 did not respond to additional scheduling requests or additional requests for information for the lab task, 3 reported stomach discomfort at a severe level and were removed).
Groups:
- Naltrexone First, Then Placebo: Participants took 4 doses of naltrexone over 4 days (25mg/day for days 1 and 2, 50mg/day for days 3 and 4) followed by a 10-day washout period and finally, 4 matched placebo pills for another 4 days.
- Placebo First, Then Naltrexone: Participants took 4 placebo pills over 4 days (one pill a day), followed by a 10-day washout period, followed by 4 naltrexone pills for 4 days (25 mg on days 1 and 2, 50mg on days 3 and 4)
Period: First Intervention
Arm/Group | Naltrexone First, Then Placebo | Placebo First, Then Naltrexone
Started | 19 | 15
Completed | 16 | 15
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Washout Period of 10 Days
Arm/Group | Naltrexone First, Then Placebo | Placebo First, Then Naltrexone
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Naltrexone First, Then Placebo | Placebo First, Then Naltrexone
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone First and Placebo First: Includes groups randomized to receive naltrexone first and placebo first.
Arm/Group | Naltrexone First and Placebo First
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.55 (3.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Self-reported Feelings of Connection During Naltrexone (vs. Placebo)
Description: Participants will read positive, loving messages from friends and family members and then rate their feelings of connection (how connected, touched, and warm they felt, α = .93, averaged to create a measure of feelings of social connection). Ratings were made on a 1-7 scale anchored by "not at all" and "very." Higher numbers indicate greater feelings of connection in response to reading the loving messages.
Time Frame: participants will report on their feelings of connection during two separate lab visits, on day 4 of each drug assignment
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Naltrexone: Participants will take 4 doses of naltrexone over 4 days (25mg/day for days 1 and 2, 50mg/day for days 3 and 4) as well as 4 matched placebo pills for a total of 8 days. Capsules will be packaged into blister packs.
  Participants will be asked to take the first drug, either naltrexone or placebo, once a day for three days prior to the first experimental session and when they arrive at the lab for the experimental procedure . After the first session, participants will take the second study drug for three days prior to the second experimental session and when they arrive for the second experimental procedure.
  Naltrexone
- Placebo: Participants will take 4 doses of naltrexone over 4 days (25mg/day for days 1 and 2, 50mg/day for days 3 and 4) as well as 4 matched placebo pills for a total of 8 days. Capsules will be packaged into blister packs.
  Participants will be asked to take the first drug, either naltrexone or placebo, once a day for three days prior to the first experimental session and when they arrive at the lab for the experimental procedure . After the first session, participants will take the second study drug for three days prior to the second experimental session and when they arrive for the second experimental procedure.
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 31 | 31
units on a scale | 5.92 (.189) | 6.47 (.183)

2. Secondary Outcome: Daily Self-reported Feelings of Social Connection
Description: For 8 days (4 while on placebo, 4 while on naltrexone), participants were asked to think back to the last 24 hours and respond to how disconnected they felt ("I felt out of touch and disconnected from others"). Ratings were made on a 1-7 scale anchored by 'strongly disagree' and 'strongly agree.' For ease of interpretation, feelings of disconnection were reverse-coded to measure daily feelings of social connection. Thus higher numbers indicate greater feelings of connection. Responses were averaged across the 4 days that participants were on each study drug (4 while on placebo, 4 while on naltrexone).
Time Frame: end of day for 8 days
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 31 | 31
units on a scale | 5.68 (0.29) | 6.26 (0.22)

3. Other Pre Specified Outcome: Self-reported Physical Symptoms
Description: At the end of each day while on a study drug (4 days when on naltrexone and 4 days when on placebo) participants reported on their physical symptoms (headaches, dizziness/faintness, nausea, appetite increase/decrease) on a 0 (no symptoms) to 4 (very severe) scale.
  Responses were averaged across study drug to evaluate a single outcome for days when participants were on naltrexone and a single outcome for days when participants were on placebo.
Time Frame: once a day for 8 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 31 | 31
units on a scale | .391 (.039) | .101 (.070)

ADVERSE EVENTS:
Time Frame: naltrexone administered once daily for 4 days (25mg for days 1 and 2, 50mg for days 3 and 4) placebo administered once daily for 4 days
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 3/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=34) | Placebo (N=34)
stomach discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No